CLINICAL TRIAL: NCT01061658
Title: Phase I/II, Randomized, Double-blind, Placebo-controlled, Dosage Selection (10e5.5 or 10e6.25 FFU of Each Constituent Serotype Per 0.5 mL) Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 3-dose Series of Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV] Administered to Healthy Indian Infants
Brief Title: Safety and Immunogenicity Study of the Tetravalent Rotavirus Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: Head, Research and Development, Shantha Biotechnics Limited, Hyderabad, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SBL/BRV-TV/Form1/PhI/2009/0100
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Rotavirus Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine - High dosage (Experimental)
  Interventions: Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine
- Vaccine - Lower dosage (Experimental)
  Interventions: Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine — Higher dosage of vaccine
  Arms: Vaccine - High dosage
Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine — Lower dosage of vaccine
  Arms: Vaccine - Lower dosage
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A double blind placebo controlled Phase I/II study to evaluate the safety and immunogenicity of the Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV]in Indian infants. The study would be carried out in 90 healthy infants. Three doses of the rotavirus vaccine or placebo would be administered orally to each infant at 6-8, 10-12 and 14-16 weeks of age. The rotavirus vaccine would be administered at one of the two planned virus concentrations (10e5.5 or 10e6.25 FFU of each constituent serotype per 0.5 ml). Each administration of the vaccine/placebo would be preceded by oral administration of 2.0 mL of antacid.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6-8 weeks of age at time of enrollment of either sex;
* Born after a gestational period of 36-42 weeks with birth weight ≥2 kg;
* Father, mother or other legally acceptable representative (guardian) properly informed about the study and having signed the informed consent form (ICF). In case of father, mother or other legally acceptable representative (guardian) being unable to read or write, having had the ICF explained to them in the presence of a study independent witness and the witness having signed the ICF;
* Parent or guardian available for the entire period of the study and reachable by study staff for post-vaccination follow-up.

Exclusion Criteria:

* History of congenital abdominal disorders, intussusception, or abdominal surgery;
* Known or suspected impairment of immunological function;
* Known hypersensitivity to any component of the rotavirus vaccine;
* Prior receipt of any rotavirus vaccine;
* Fever, with axillary temperature ≥38.1oC (≥100.5oF); measured by study staff.
* History of known rotavirus disease, chronic diarrhea, or failure to thrive;
* Baseline level of ALT or AST >2.5 times the upper limit of normal;
* Clinical evidence of active gastrointestinal illness (infants with GERD can participate in the study so long as this condition is well controlled with or without medication);
* Receipt of any IM, oral, or IV corticosteroid treatment in the past 30 days (infants on inhaled steroids may be permitted to participate in the study);
* Infants residing in a household with an immuno-compromised person (e.g., individuals with a congenital immunodeficiency, HIV infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure, nephrotic syndrome, organ or bone marrow transplantation, or those receiving immunosuppressive chemotherapy including long-term systemic corticosteroids);
* Infants suspected to be HIV, HBV or HCV positive from the available clinical history or born to mothers known to be HIV, HBV or HCV positive.
* Prior receipt of a blood transfusion or blood products, including immunoglobulins;
* Any infants who cannot be adequately followed for safety by a home visit;
* Any conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Parent/s or guardian of subject unable to maintain diary card

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The frequency, severity, and causality of Reactogenicity Events and other Adverse Events. | After each dose and upto 28 days after third dose

SECONDARY OUTCOMES:
The Seroconversion rate, Sero-response rate and the GMT of serum IgA antibody against rotavirus. | After each dose and upto 28 days after third dose
The frequency and duration of post-vaccination shedding of vaccine rotavirus in stool samples | After each dose and upto 7 days after third dose

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India